CLINICAL TRIAL: NCT02049866
Title: Denosumab for Prevention of Post-Teriparatide Bone Loss in Premenopausal Women With Idiopathic Osteoporosis (IOP)
Brief Title: Denosumab for Prevention of Post-Teriparatide Bone Loss in Premenopausal Women With IOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elizabeth Shane (Other)
Collaborators: Creighton University (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Shane, Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAN0161; 1R01FD005114-01A2 (FDA)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-10

CONDITIONS: Adult Idiopathic Generalized Osteoporosis
Keywords: osteoporosis; premenopausal; denosumab; idiopathic; Idiopathic Osteoporosis in Premenopausal Women
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Denosumab (Experimental): Denosumab 60mg, administered every 6 months by subcutaneous injection for 36 months.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Denosumab 60mg, administered every 6 months by subcutaneous injection for 36 months
  Other Names: Prolia; Xgeva

SUMMARY:
The purpose of this research study is to evaluate antiresorptive therapy with denosumab (Prolia) for prevention of bone loss after stopping teriparatide (TPTD) in premenopausal women with idiopathic osteoporosis.

Premenopausal women who have received TPTD in the FDA Orphan Diseases Program-funded trial, "A Phase 2 Study of Teriparatide for the Treatment of Idiopathic Osteoporosis in Premenopausal Women" (NCT01440803) may be eligible to participate in the current study, a 36-month open-label pilot study of denosumab (Prolia®, 60mg subcutaneous (SC) every 6 months).

The goals of the study are to estimate the effects of denosumab on central and peripheral, as well as trabecular and cortical, bone mass and microstructure and to obtain preliminary data to inform the design of a future randomized study. This study presents the first opportunity to study the effects of denosumab after TPTD in this unique and severely affected group of young women.

Funding Source: FDA Office of Orphan Products Development (OOPD).

DETAILED DESCRIPTION:
Osteoporosis in premenopausal women with normal menstrual function and no specific cause is termed idiopathic osteoporosis (IOP). IOP is a rare disease with an estimated prevalence of <200,000 affected premenopausal women in the United States.

Denosumab, a potent inhibitor of osteoclast-mediated bone resorption, leads to continuous gains in both trabecular and cortical bone mineral density (BMD). Moreover, denosumab is not retained in the skeleton, and may thus be preferable for use in young women who may be contemplating future pregnancies. The investigators hypothesize that denosumab, initiated after completion of two years of TPTD, will maintain or improve central and peripheral areal and volumetric BMD, microstructure and stiffness in premenopausal women with IOP.

ELIGIBILITY:
Inclusion Criteria:

* All women completing NCT01440803 who remain without a disease or medication that causes osteoporosis will be offered enrollment into this study.
* (Premenopausal status is no longer be required for entry.)

Exclusion Criteria:

* Renal insufficiency or liver disease: Creatinine, transaminase (AST)/alanine transaminase (ALT) above upper limit of normal
* Vitamin D deficiency: 25-hydroxyvitamin D (25-OHD) <30 ng/mL
* Pregnancy: urine pregnancy test must be negative

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shane, MD, Principal Investigator — Columbia University; Adi Cohen, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Creighton University, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shane E, Shiau S, Recker RR, Lappe JM, Agarwal S, Kamanda-Kosseh M, Bucovsky M, Stubby J, Cohen A. Denosumab After Teriparatide in Premenopausal Women With Idiopathic Osteoporosis. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1528-e1540. doi: 10.1210/clinem/dgab850. PMID 34849989
- See also: Columbia University, Dept of Medicine, Division of Endocrinology website — http://columbiamedicine.org/divisions/Endo/index.shtml

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Denosumab
Started | 33
Completed | 32
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Denosumab
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Lumbar Spine Areal BMD by DXA
Description: Bone mineral density (BMD) will be measured with dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and 12 months
Population: 33 participants completed baseline but 1 participant withdrew from the study before the 12 month visit.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Denosumab
Number analyzed (Participants) | 32
percentage of change | 5.2 (2.6)

2. Secondary Outcome: Percent Change in Lumbar Spine Areal BMD by DXA at 24 Months
Description: Bone mineral density (BMD) will be measured with dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Denosumab
Number analyzed (Participants) | 29
percentage of change | 6.9 (2.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 year (from baseline to 12 month study participation).
Arm/Group | Denosumab
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 26/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Denosumab (N=33)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) — Nonvertebral fragility fracture
Redness (Surgical and medical procedures) | 2 (2) — Redness at injection site reaction
Pain (Surgical and medical procedures) | 9 (9) — Injection site reaction
Urinary tract infection (Infections and infestations) | 12 (12)
Ear infection (Infections and infestations) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hair loss (Skin and subcutaneous tissue disorders) | 3 (3)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 4 (4)
Numbness and/or tingling (Nervous system disorders) | 6 (6)
Nausea and vomiting (Gastrointestinal disorders) | 2 (2)
Pain in thighs, hips, or groin (Musculoskeletal and connective tissue disorders) | 11 (11)
Cold (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Low Energy (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT02049866/Prot_SAP_000.pdf